CLINICAL TRIAL: NCT00263549
Title: Multicenter Study for Evaluation of Efficacy and Safety of Perennial Specific Immunotherapy With a Depot House Dust Mite Allergen Extract (D. Pteronyssinus 100%) in Patients With House Dust Mite Sensitivity
Brief Title: Safety and Efficacy of House Dust Mite Allergen Extract in the Treatment of Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Al0201NH
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: House Dust Mite Allergy
Keywords: House dust mite,; Allergy
MeSH Terms: conditions — Dust Mite Allergy; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: House dust mite Novo Helisen Depot

SUMMARY:
The trial is performed to assess efficacy and safety of Novo-Helisen Depot in allergic Rhinoconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test to house dust mite,
* Positive RAST test to house dust mite,
* Positive provocation test result to house dust mite,

Exclusion Criteria:

* Serious chronic diseases,
* Other perennial allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2002-09; Primary Completion 2005-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M.D., Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de